CLINICAL TRIAL: NCT02904746
Title: A Brief, Trauma-Informed Intervention to Increase Treatment Engagement Among Individuals Referred for Post-Crisis Mental Health Services
Brief Title: Intervention to Increase Treatment Engagement Among Individuals Referred for Post-Crisis Mental Health Services
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to successfully recruit participants using current study design.
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Natalie Mota, Assistant Professor/Staff Psychologist, University of Manitoba
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H2016:124
Record Dates: First submitted 2016-09-07; First posted 2016-09-19 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2017-05

CONDITIONS: Mental Health Crisis
Keywords: follow-up; mental health appointment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Participants receiving the Make It! intervention
  Interventions: Behavioral: Make It!
- Control (No Intervention): Care as usual

INTERVENTIONS:
Behavioral: Make It! — The Make It! motivational enhancement intervention has been informed by Motivational Interviewing principles, a method that has widely demonstrated effectiveness in increasing a number of positive behavior changes, including appointment adherence. Make It! consists of a 10-15 minute intervention with 5 components: Common reactions to stressors that this exposure can lead to a range of reactions, pros and cons of attending the Information Class, visualization of the Information Class, expression of confidence that the client can progress towards change, and reiteration of main information.
  Arms: Intervention

SUMMARY:
This study will evaluate the preliminary effectiveness of Make It!, a single 15-minute intervention aimed at increasing attendance to a follow-up appointment for psychological services (i.e., an information class) among clients accessing walk-in services at a mental health crisis response centre. As a secondary aim, we will examine the demographic correlates, presenting problems, and symptom correlates of clients who do and do not attend follow-up services.

DETAILED DESCRIPTION:
The current study will employ a quasi-experimental design whereby several frontline clinicians at a mental health crisis response will be trained to deliver the Make It! intervention and the others will not. An attempt will be made to train staff who commonly share work days or shifts in order to avoid details of the active intervention reaching clinicians who continue to deliver treatment as usual. For the duration of the study period, clinicians trained in Make It! will be instructed to use the intervention as their standard of care with all of the clients they assess whom are subsequently referred to the Information Class. The remaining clinicians will continue to use treatment as usual.

During a 90 minute workshop, Make It! will be introduced and modeled by the Principal Investigator (PI). Make It! consists of a 10-15 minute intervention with 5 components: 1) Acknowledgement that the client has experienced distressing events and/or very stressful situations, and that this exposure can lead to a range of reactions, 2) Client-generated, clinician-assisted, pros and cons of attending the Information Class, 3) Detailed visualization of the First Information in order to reduce anxiety about what to expect, 4) Expression of confidence that the client can begin progress towards the changes they want to make, 5) Reiteration of main information and appointment card given. Each clinician trained will be observed administering the intervention to a co-worker, with fidelity checks being implemented throughout the study period. These fidelity checks will be implemented by the PI, who will occasionally and sporadically observe the clinicians administer the intervention through a one-way mirror, with the verbal consent of the participant and the clinician.

All clients accessing the walk-in service at the crisis response centre currently receive a mental health assessment by a staff clinician. Throughout the course of the assessment, if the clinician perceives that the client may benefit from follow-up psychological services, he or she provides the client with an appointment date and time for the next available Information Class. The Information Class is a group appointment, and its purpose is to provide information about the services offered at the centre. It serves as the entryway into follow-up services such as cognitive behavioral therapy classes for mood and anxiety symptoms or dialectical behavioral therapy-informed classes. Walk-in clients who receive an appointment for this Information Class typically are given an appointment date that is within 1-2 weeks of their walk-in visit.

Once the clinician makes a decision to refer a client to an Information Class, the clinician will contact the study coordinator. The study coordinator or research volunteer will come into the interview room while the clinician steps out, will explain the study to the participant, and will obtain informed consent. In the event that a potential participant requires more time to consider whether he or she wants to consent to study participation, the individual will be provided with the contact information of the study coordinator in order to be able to consent at a later date. The study coordinator or research volunteer will also ask the participant to complete some brief questionnaires at this time assessing barriers to seeking mental health care and stages of change.

The study coordinator or research volunteer will then leave and the clinician will return to the interview room. If the clinician has not been trained in Make It!, he/she will proceed with care as usual. This condition involves providing the client with detailed information about the upcoming Information Class. If the clinician has been trained in Make It!, then the intervention will proceed at this time.

A few days before the client's Information Class, a reminder call is made by an administrative assistant at the centre. When the administrative assistant is unable to reach the client, she leaves a brief message, if possible to do so.

On the day of the Information Class, attendance will be taken. Clients sit in a classroom setting and complete a package of questionnaires. Those participants enrolled in the study will complete the Life Events Checklist-5, the University of Rhode Island Change Assessment, and an open-ended question assessing barriers to care, in addition to 5 questionnaires assessing a range of mental health symptoms that are already administered at the Information Class for clinical purposes. After the Information Class, clients have the opportunity to meet individually for 5-10 minutes with a staff member in order to discuss their treatment needs and preferences, and to connect them with subsequent services. If the client is a participant in the study, the staff member will provide them with a debriefing document that also contains the PI's contact information should they have any additional questions, comments, or concerns. This concludes the client's participation in the study.

For study participants who do not attend the Information Class, the questionnaires administered at the Information Class will be mailed to the participant along with a standard Information Class "no show" letter and the study's debriefing document. Participants will be encouraged to complete the questionnaires and return them in the self-addressed stamped envelope to the PI. This will represent the end of the participant's role in the study.

If a participant calls in advance of the Information Class to reschedule their Class date, or if they inform the administrative assistant that they wish to reschedule when she makes the reminder call, the participant will continued to be considered a participant until their rescheduled appointment.

ELIGIBILITY:
Criteria for being referred to the crisis centre's Information Class and thus, for participation in the study are:

* presenting to the walk-in service with a mental health-related crisis (e.g., difficulty coping with acute stressors, suicidality),
* a willingness by the client to participate in class-based or group interventions,
* the ability to attend and have transportation to services during daytime hours,
* the client is not better served by another service for their presenting problem (e.g., Addictions Foundation of Manitoba when alcohol or substance is primary),
* the client is literate and will be able to understand and benefit from attending class-based or group psychotherapy interventions, and
* the client is not being admitted to the Crisis Stabilization Unit or hospital (i.e., is not at imminent risk of harming themselves or others).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Attendance status to Information Class | 1-2 weeks post enrollment in study

SECONDARY OUTCOMES:
University of Rhode Island Change Assessment (URICA) | Immediately following study enrolment and 1-2 weeks post enrollment in study
Open-ended question regarding barriers to pursuing mental health services | Immediately following study enrollment and 1-2 weeks post enrollment in study (at Information Class)
Patient Health Questionnaire-9 (PHQ-9) | 1-2 weeks post enrollment in study (at Information Class)
Generalized Anxiety Disorder Questionnaire (GAD-7) | 1-2 weeks post enrollment in study (at Information Class)
Posttraumatic Stress Disorder Checklist-5 (PCL-5) | 1-2 weeks post enrollment in study (at Information Class)
Diagnostic and Statistical Manual of Mental Disorders (DSM-5) Cross-cutting Measure | 1-2 weeks post enrollment in study (at Information Class)
Difficulties in Emotion Regulation Scale (DERS) | 1-2 weeks post enrollment in study (at Information Class)
Age | To be extracted from client's medical record immediately following enrolment in study
Gender | To be extracted from client's medical record immediately following enrolment in study
Marital status | To be extracted from client's medical record immediately following enrolment in study
Employment status | To be extracted from client's medical record immediately following enrolment in study
Presenting problem at walk-in visit to crisis centre | To be extracted from client's medical record immediately following enrolment in study

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Mota, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Crisis Response Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No